CLINICAL TRIAL: NCT01282801
Title: Randomized, 2-way Crossover, Bioequivalence Study of Venlafaxine Hydrochloride 150 mg Extended-Release Capsules and Effexor® XR 150 mg Extended-Release Capsules Administered as 1 x 150 mg Extended-Release Capsules in Healthy Subjects Under Fed Conditions.
Brief Title: Venlafaxine Hydrochloride 150 mg Extended-Release Capsules Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, Teva Pharmaceuticals, USA
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 02205
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Results first posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Venlafaxine Hydrochloride

ARMS (2):
- Investigational Test Product (Experimental): Venlafaxine Hydrochloride 150 mg Extended-Release Capsules
  Interventions: Drug: Venlafaxine Hydrochloride
- Reference Listed Drug (Active Comparator): Effexor® XR 150 mg Extended-Release Capsules
  Interventions: Drug: Effexor® XR

INTERVENTIONS:
Drug: Venlafaxine Hydrochloride — 150 mg Extended-Release Capsule
  Arms: Investigational Test Product
Drug: Effexor® XR — 150 mg Extended-Release Capsule
  Other Names: Venlafaxine Hydrochloride (generic name)
  Arms: Reference Listed Drug

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of venlafaxine hydrochloride 150 mg extended-release capsules (test) versus Effexor® XR (reference) administered as 1 x 150 mg extended-release capsule under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Members of the community at large.
* Subjects will be females and/or males, non-smokers, 18 years of age and older.
* Female subjects will be post-menopausal or surgically sterilized.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any history or presence of significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* History or presence of any clinically significant gastrointestinal pathology, unresolved gastrointestinal symptoms, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Subjects with raised intra-ocular pressure or at risk of acute narrow angle glaucoma.
* Subjects predisposed to bleeding of the skin and mucous membrane.
* Subjects with a history of seizures.
* Any reason which, in the opinion of the medical sub-investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities at screening.
* Subjects with BMI > 30.0.
* History of significant alcohol abuse within six months of screening visit or any indication of the regular use of more than fourteen units of alcohol per week (1 unit equals 150 mL of wine, 360 mL of beer, or 45 mL of alcohol 45%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (cocaine, PCP, crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction, or special diet that, in the opinion of the medical sub-investigator, contraindicates the subject's participation in the study.
* History of allergic reactions to venlafaxine hydrochloride.
* History of allergic reactions to heparin.
* Use of any drugs know to induce or inhibit hepatic drug metabolism, use of an investigational drug, or participation in an investigational study within 30 days prior to administration of the study medication.
* Use of prescription medication within 14 days prior to administration of the study medication or over-the-counter products within 7 days prior to the administration of study medication, except for topical products without systemic absorption.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of the study medication.
* Donation of plasma (500 mL) within 7 days of Period I dosing. Donation or loss of whole blood prior to administration of the study medication as follows:

  * less than 300 mL of whole blood within 30 days or
  * 300 mL to 500 mL of whole blood within 45 days or
  * more than 500 mL of whole blood within 56 days.
* Positive alcohol breath test at screening.
* Subjects who have used tobacco in any form within the 90 days preceding study drug administration.
* Subjects who have consumed food or beverages containing grapefruit within 7 days prior to administration of the study medication.
* Intolerance to venipunctures.
* Additional exclusion criteria for females only:

  * Breastfeeding subjects.
  * Positive urine pregnancy test at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-09; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Velafaxine Hydrochloride (Test) First: 150 mg Venlafaxine Hydrochloride Extended-Release Capsules test product dosed in first period followed by 150 mg Effexor® XR Capsules reference product dosed in the second period.
- Effexor® XR (Reference) First: 150 mg Effexor® XR Extended-Release Capsules reference product dosed in first period followed by 150 mg Venlafaxine Hydrochloride Extended-Release Capsules test product dosed in the second period.
Period: First Intervention
Arm/Group | Velafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Velafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Velafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First
Started | 9 | 9
Completed | 9 | 8
Not Completed | 0 | 1
Not completed — Emesis During Critical Breakfast | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Velafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 5 | 8 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Venlafaxine.
Description: Bioequivalence based on Venlafaxine Cmax (maximum observed concentration of drug substance in plasma).
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Velafaxine Hydrochloride (Test): 150 mg Venlafaxine Hydrochloride Extended-Release Capsules test product dosed in either period.
- Effexor® XR (Reference): 150 mg Effexor® XR Extended-Release Capsules reference product dosed in either period.
Arm/Group | Velafaxine Hydrochloride (Test) | Effexor® XR (Reference)
Number analyzed (Participants) | 17 | 17
ng/mL | 81.84 (37.59) | 93.50 (37.73)

2. Primary Outcome: AUC0-t of Venlafaxine.
Description: Bioequivalence based on Venlafaxine AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration).
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Velafaxine Hydrochloride (Test) | Effexor® XR (Reference)
Number analyzed (Participants) | 17 | 17
ng*h/mL | 1358.37 (766.51) | 1383.57 (769.22)

3. Primary Outcome: AUC0-inf of Venlafaxine.
Description: Bioequivalence based on Venlafaxine AUC0-inf (area under the concentration-time curve from time zero to infinity).
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Velafaxine Hydrochloride (Test) | Effexor® XR (Reference)
Number analyzed (Participants) | 17 | 17
ng*h/mL | 1596.83 (902.89) | 1605.29 (910.77)

4. Secondary Outcome: Cmax of O-Desmethylvenlafaxine.
Description: Informational comparison of Cmax values for the metabolite O-Desmethylvenlafaxine.
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Velafaxine Hydrochloride (Test) | Effexor® XR (Reference)
Number analyzed (Participants) | 17 | 17
ng/mL | 227.02 (48.08) | 236.21 (57.37)

5. Secondary Outcome: AUC0-t of O-Desmethylvenlafaxine.
Description: Informational comparison of AUC0-t values for the metabolite O-Desmethylvenlafaxine.
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Velafaxine Hydrochloride (Test) | Effexor® XR (Reference)
Number analyzed (Participants) | 17 | 17
ng*h/mL | 5591.56 (1412.83) | 5748.06 (1578.70)

6. Secondary Outcome: AUC0-inf of O-Desmethylvenlafaxine.
Description: Informational comparison of AUC0-inf values for the metabolite O-Desmethylvenlafaxine.
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Velafaxine Hydrochloride (Test) | Effexor® XR (Reference)
Number analyzed (Participants) | 17 | 17
ng*h/mL | 7945.58 (2636.77) | 8102.12 (2769.50)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 2 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Velafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 12/18 | 14/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velafaxine Hydrochloride (Test) First (N=18) | Effexor® XR (Reference) First (N=18)
Sore Throat (General disorders) | 1 (1) | 0 (0)
Runny Nose (General disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 4 (4) | 8 (9)
Drowsiness (General disorders) | 1 (1) | 3 (3)
Vomiting (General disorders) | 0 (0) | 1 (1)
High Blood Pressure (General disorders) | 5 (6) | 4 (4)
Loose Stools (General disorders) | 1 (1) | 1 (1)
Dizziness (General disorders) | 1 (1) | 1 (1)
Difficulty Swallowing (General disorders) | 0 (0) | 1 (1)
Tremors (General disorders) | 0 (0) | 1 (1)
Redness of Arm (General disorders) | 1 (1) | 0 (0)
Pain at Catheter Site (General disorders) | 1 (1) | 0 (0)
Hot Flushes (General disorders) | 1 (1) | 0 (0)
Swelling of Hand (General disorders) | 1 (1) | 0 (0)
Swollen Arm (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1)
Bruising of Hand (General disorders) | 1 (1) | 0 (0)
Leukocytes in Urine (General disorders) | 0 (0) | 1 (1)
Flatulence (General disorders) | 1 (1) | 1 (1)
Difficulty Sleeping (General disorders) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 1 (1)
Delayed Ejaculation (General disorders) | 1 (1) | 1 (1)
Protein in Urine (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.